CLINICAL TRIAL: NCT06804811
Title: A Phase 3, Randomized, Double-Blind, Efficacy, and Safety Study of Ruxolitinib Cream in Children (6 to < 12 Years Old) With Nonsegmental Vitiligo
Brief Title: A Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Children (6 to < 12 Years Old) With Nonsegmental Vitiligo
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB18424-309; 2024-513171-41-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: NonSegmental Vitiligo
Keywords: NonSegmental Vitiligo; pediatric

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ruxolitinib 0.75 % Cream (Experimental): Participants received ruxolitinib 0.75% cream, applied topically to the affected area as defined in the protocol.
  Interventions: Drug: Ruxolitinib Cream
- Ruxolitinib 1.5 % Cream (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected area as defined in the protocol.
  Interventions: Drug: Ruxolitinib Cream
- Vehicle Cream (Placebo Comparator): Participants received vehicle cream, applied topically to the affected area as defined by the protocol.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream applied topically to the affected area as a thin film twice daily.
  Other Names: INCB018424 Phosphate Cream
  Arms: Ruxolitinib 0.75 % Cream; Ruxolitinib 1.5 % Cream
Drug: Vehicle Cream — Matching vehicle cream applied topically to the affected area as a thin film twice daily.
  Arms: Vehicle Cream

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib cream in children (6 to < 12 years old) with nonsegmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to < 12 years at the time of signing the ICF.
* Clinical diagnosis of nonsegmental vitiligo with depigmented area including ≥ 0.5% BSA on the face, ≥ 0.5 F-VASI, ≥ 3% BSA on nonfacial areas, ≥ 3 T-VASI.
* Total body vitiligo area does not exceed 10% BSA.
* Pigmented hair within some of the areas of vitiligo on the face.
* Must agree to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit.
* For sexually active participants (except participants who are prepubescent) willingness to avoid pregnancy or fathering a child as defined in the protocol.

Exclusion Criteria:

* Diagnosis of other forms of vitiligo (eg, segmental).
* Other differential diagnosis of vitiligo or other skin depigmentation disorders (eg, piebaldism, pityriasis alba, leprosy, postinflammatory hypopigmentation, progressive macule hypomelanosis, nevus anemicus, chemical leukoderma, and tinea versicolor).
* Any other skin disease that, in the opinion of the investigator, would interfere with the study drug application or study assessments.
* Prior or current use of depigmentation treatments (eg, monobenzone).
* Concurrent conditions and history of protocol-defined diseases
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including application of study cream and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Use of protocol-defined treatments within the indicated washout period before baseline.
* History of treatment failure with any systemic or topical JAK inhibitor for vitiligo or any other inflammatory condition.
* Protocol-defined clinically significant abnormal laboratory values at screening.
* BMI-for-age < 5th percentile or ≥ 85th percentile according to the CDC BMI Percentile Calculator for Child and Teen.
* Pregnant or lactating participants or those considering pregnancy during the period of their study participation.
* In the opinion of the investigator, unable or unlikely to comply with the application schedule and study evaluations.
* Living with anyone participating in any current Incyte-sponsored ruxolitinib cream study.
* Employees of the sponsor or investigator or are otherwise dependents of them.
* Known allergy or reaction to any component of the study cream formulation.
* The following participants are excluded in France: vulnerable populations according to article L.1121-6 of the French Public Health Code and adults under legal protection, or who are unable to express their consent per article L.1121-8 of the French Public Health Code, not affiliated to a social security per article L.1121-8-1 of the French Public Health code.
* In the EU, participants considered incapacitated according to EU CTR No. 536/2014 Articles 2 and 31.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving a ≥ 75% Improvement From Baseline in the Facial Vitiligo Area Scoring Index (F-VASI75) | Week 24
  ≥75% improvement in facial Vitiligo Area Scoring Index.

SECONDARY OUTCOMES:
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI50) | Week 24
  ≥50% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI90) | Week 24
  ≥90% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving a ≥ 50% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) | Week 24
  ≥50% improvement in total body Vitiligo Area Scoring Index.
Percentage change from baseline in F-BSA | Week 24
  Facial body surface area (F-BSA) takes into account the facial depigmented areas as a percentage of the total body area.
Number of Treatment Emergent Adverse Events (TEAEs) | Up to Week 52 and 30 days
  TEAE defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Proportion of participants achieving a Vitiligo Noticeability Scale (VNS) score of 4 (a lot less noticeable) or 5 (no longer noticeable) | Week 24 and Week 52
  The VNS is a patient-reported measure of vitiligo treatment success that has a 5-point scale.
Proportion of participants in each category for the color-matching question | Week 24 and Week 52
  The color-matching question is a patient-reported measure of vitiligo treatment success that has a 5-point scale.
Proportion of participants who report facial assessment of Patient Global Impression of Change-Vitiligo (F-PaGIC-V) of very much improved or much improved | Week 24 and Week 52
  The F-PaGIC-V is an assessment of improvement by the participant that has a 7-point scale.
Proportion of participants who report total body assessment of Patient Global Impression of Change-Vitiligo (T-PaGIC-V) of very much improved or much improved | Week 24 and Week 52
  The T-PaGIC-V is an assessment of improvement by the participant that has a 7-point scale.
Change from baseline in Psychosocial Impact Questionnaire for Pediatric Patients Who Have Nonsegmental Vitiligo (VIT-PIQ) | Week 24 and Week 52
  The VIT-PIQ is a 17-item questionnaire to assess Quality of Life (QOL) of children with vitiligo.
Change from baseline in Children's Dermatology Life Quality Index (CDLQI) | Week 24 and Week 52
  The CDLQI is the youth/children's version of the Dermatology Life Quality Index.
Change from baseline in Patient Global Impression of Bother - Vitiligo (PGIB-V) | Week 24 and Week 52
  The PGIB-V is a single question with an 11-point scale ("not at all" to "a whole lot") to assess the participant's level of bother because of their vitiligo.
Mean satisfaction score | Week 24 and Week 52
  The treatment satisfaction tool is a fit-for-purpose questionnaire to assess treatment satisfaction in children with nonsegmental vitiligo.
Pharmacokinetic (PK) of Ruxolitinib: Trough concentrations | Weeks 6, 24, 30 and 52
  Trough is defined as the concentration reached by a drug immediately before the next dose is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (86):
- Argentina (8):
  - Psoriahue, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto de Neumonologia Y Dermatologia, Buenos Aires
  - Consultorios Medicos Dr. Doreski, Buenos Aires
  - Derma Internacional S.A., Buenos Aires
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Hospital Universitario Austral, Pilar
  - Hospital Del Nino Jesus, San Miguel de Tucumán
- Austria (2):
  - Universitaetsklinikum Graz, Graz
  - Medical University Innsbruck, Innsbruck
- Belgium (4):
  - Hopital Universitaire de Bruxelles (Academisch Ziekenhuis Brussel), Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Universite Catholique de Louvain (Ucl) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Bulgaria (8):
  - Medical Center Asklepii Ood, Dupnitsa
  - Mhat Dr. Tota Venkova Ad, Gabrovo
  - Medical Center Medkonsult Pleven Ood, Pleven
  - Medical Center Unimed Eood, Sevlievo
  - Umhat Aleksandrovska, Sofia
  - 28 Diagnostic and Consultative Center, Sofia
  - Mc Euroderma Clinic, Sofia
  - Diagnostic Consultation Center Xx - Sofia Eood, Sofia
- Denmark (2):
  - Sanos Clinic, Gandrup
  - Herlev and Gentofte Hospital, Hellerup
- France (10):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Universitaire (Chu) de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Hospices Civils de Lyon (Hcl) - Hopital Edouard Herriot (Heh), Lyon
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hopital Hotel Dieu, Nantes
  - Centre Hospitalier Universitaire de Nice,Hopital L Archet, Nice
  - Hopital Universitaire Necker Enfants Malades, Paris
  - Polyclinique de Courlancy, Reims
  - Centre Hospitalier Universitaire (Chu) de Toulouse - Hopital Larrey, Toulouse
  - Chu Nancy, Vandœuvre-lès-Nancy
- Germany (11):
  - Charite - Universitaetsmedizin Berlin - Campus Charite Mitte (Ccm), Berlin
  - Universitaetsklinikum Der Ruhr Universitaet Bochum (Ukrub), St. Josef Hospital, Bochum
  - Drk Krankenhaus Chemnitz-Rabenstein, Chemnitz
  - Hautklinik Universitatsklinikum Erlangen, Erlangen
  - Universitaetsklinik Frankfurt, Frankfurt
  - Katholisches Kinderkrankenhaus Wilhelmstift, Hamburg
  - University Medical Center Schleswig-Holstein, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Klinikum Rechts Der Isar Der Technischen Universitaet Muenchen (Hopital Rechts Der Isar), München
  - University Hospital Muenster, Münster
- Hungary (4):
  - Clinexpert, Budapest
  - Debreceni Egyetem Klinikai Kozpon Belgyogy Klinika, Debrecen
  - University of Pecs-Clinical Center, Pécs
  - University of Szeged, Szeged
- Italy (10):
  - A.O. Policlinico Sant'Orsola Malpighi-Universita Degli Studi Di Bologna, Bologna
  - Azienda Ospedaliera Spedali Civili Di Brescia-Universita Degli Studi Di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria Policlinico Vittorio Emanuele Ospedale Gaspare Rodolico Di Catania, Catania
  - Uoc Dermatologia Ospedale Maggiore Policlinico, Fondazione Irccs Ca' Granda, Milan
  - Universita Degli Studi Di Napoli Federico Ii, Napoli
  - Azienda Ospedale Universita Di Padova, Padua
  - Fondazione Ptv Policlinico Tor Vergata, Roma
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Ircss), Roma
  - Irccs Ospedale Pediatrico Bambino Gesu, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Rome
- Amsterdam Umc Research Bv, Amsterdam, Netherlands
- Poland (10):
  - Centrum Badan Klinicznych Pi-House Sp. Z O.O., Gdansk
  - Care Clinic Sp. Z O.O., Katowice
  - Diamond Clinic Specjalistyczne Poradnie Lekarskie, Krakow
  - Dermedic Iwona Zdybska, Lublin
  - Twoja Przychodnia - Medyczne Nowa Sol, Nowa Sól
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski, Osielsko
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Uniwersytecki Szpital Kliniczny Im. Fryderyka Chopina W Rzeszowie, Rzeszów
  - Twoja Przychodnia Scm, Szczecin
  - Evimed Sp. Z O. O., Warsaw
- Portugal (3):
  - Centro Hospitalar E Universitario Coimbra, Coimbra
  - Centro Hospitalar de Lisboa Central - Hospital Santo Antonio Dos Capuchos, Lisbon
  - Hospital Geral de Santo Antonio, Porto
- Spain (6):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Sant Joan de Deu Barcelona, Esplugues de Llobregat
  - Hospital Infantil Unversitario Nino Jesus, Madrid
  - Hospital Universitario Miguel Servet de Zaragoza, Zaragoza
- United Kingdom (7):
  - Croydon University Hospital, Croydon
  - The Royal London Hospital - Barts Health Nhs Trust, London
  - Guys Hospital, London
  - Great Ormond Street Hospital For Children Nhs Foundation Trust, London
  - Queen'S Medical Centre - Nottingham University Hospitals Nhs Trust, Nottingham
  - Sheffield Childrens Hospital, Sheffield
  - Manor Hospital (Walsall) - Walsall Healthcare Nhs Trust, Walsall

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Children (6 to < 12 Years Old) With Nonsegmental Vitiligo — https://incyteclinicaltrials.com/studies/incb18424-309